CLINICAL TRIAL: NCT04076969
Title: Effect of an Integrated Educational Session on Enhancing Compliance Behavior Among Pregnant Women With Iron Deficiency Anemia
Brief Title: Integrated Educational Session and Enhancing Compliance Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Mahmoud Abdel Ghani, Assisstant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 00004025
Record Dates: First submitted 2019-08-28; First posted 2019-09-04 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Anemia; Iron-deficiency
Keywords: Iron deficiency; Moderate anemia; Compliance
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency; Iron Deficiencies; Patient Compliance

STUDY DESIGN:
Intervention Model Description: there are two groups, the study group and the control group
Who Masked: Participant
Masking Description: The pregnant women were blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Educational Session (Experimental): The anemic pregnant women in the study group received an integrated health education in one session. The educational session was steered as 40-minutes session in a personalized manner. The educational session content included; disease specific information, effect of anemia on maternal and neonatal outcome, management possibilities, the effectiveness, benefits and disadvantages of treatment options, identify diet rich with iron, false dietary habits prevent iron absorption and the balanced diet and meals.
  Interventions: Behavioral: Integrated educational session
- Routine follow up (Other): Routine follow up
  Interventions: Behavioral: Integrated educational session

INTERVENTIONS:
Behavioral: Integrated educational session — The educational session aimed to correct the pregnant women diatery habits and enhance the degree of compliance to the iron treatment and follow up instruction.

SUMMARY:
This study aimed to determine the effect of an integrated educational session on enhancing compliance behavior among pregnant women with iron deficiency anemia.The anemic pregnant women in the study group received an integrated health education in one session. While pregnant women who were allocated to the control group received the routine antenatal care and follow up.

DETAILED DESCRIPTION:
Data collection was conducted between April 2019 and December 2019.This study was grounded in the health compliance model(Heiby and Carlson, 1986) which proposed that elements of engagement between health care providers and patients involve activities that are likely to promote the development of information, produce productive emotions, and help develop the skills required to conduct health behavior. Such aspects of engagement include the healthcare provider listening to the patient's questions, engaging the patient in treatment decisions, and evaluating comprehension of the patient.

For the first interview at 24 weeks' gestation, the pregnant women were re-informed about the purpose of the study and the schedule of follow-up. The baseline data that was gathered included test of the women's Hb levels during their routine antenatal visit, socio-demographic characteristics, and obstetric history. Three follow-up examinations were planned for pregnant women in both study and control groups at weeks 28, 32 and 36 of gestation. In the study group, pregnant women with anemia obtained an integrated health education in one session. The educational session was conducted by the principle investigator (PI) and was steered as 40-minutes session and provided individually to every participating woman. The content of the educational session included; disease specific knowledge, impact of anemia on maternal and neonatal outcomes, management opportunities, effectiveness, advantages and draw¬backs of treatment choices, iron-rich diet recognition, false eating patterns stopping iron absorption, and healthy diet. The PI has adopted the medical recommendations based on dietary guidelines for pregnancy(WHO, 2012). The pregnant women were given a chance to ask questions related to the session and its content. Furthermore, women were educated in recording all food and drink consumed inside and outside of the home, i.e. each meal/dish they got during the reporting duration of their diary, 24 hours of recall for seven days. They were also asked to report the exact portion size of the food by normal household measurements (e.g. plates, pots, cups, spoons, and glasses) or by kitchen scale. Additionally, each woman was advised to select the easiest way to remind her of her vitamin time.

The pregnant women received an educational brochure at the end of the educational session which included all the information given in that session written in Arabic language. The literature-based educational brochure material was reviewed by three experts in the field of maternity nursing prior to the distribution. Each pregnant woman in both study and control groups was evaluated twice at 28 and 36 weeks' gestation for total dietary iron. The dietary iron intake recorded by women has been calculated using the IRONIC-FFQ and revised, when needed, by dietitian who was not involved in the study. In addition, the degree of the women's adherence to medication was measured by counting the total numbers of pills consumed between two scheduled appointments. For antenatal follow-up appointments for all women in the study and the control groups, phone calls were given monthly and women were reminded to record the iron intake diary seven days before their appointment. The participants returned their supplementary bottles with any unused capsules to the PI during their monthly visits to the antenatal clinic. Adherence to the supplementation scheme was determined based on the number of capsules left in the package after each return visit; adherence (percent)=[30-number of pills left in the package/number of days between the date of dispensation and the date of return]100. The equation was adopted based on the method used in(Cogswell et al., 2003).

At the last data collection occasion at gestation week 36, the medication adherence scale was inserted along with check of Hb levels for all participating women. Pregnant women who were allocated to the control group received the routine antenatal care and follow-up, but no educational sessions or materials were provided to them

Primary Outcome:

Compliance degree

Secondary Outcome:

Iron food intake/mg, the hemoglobin level & ferritin levels

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Primiparous
* Singleton pregnancy
* Literate

  *± 24 weeks gestation
* Diagnosed moderate anemia
* With normal BMI on booking (i.e. 24-25)

Exclusion Criteria:

* Pregnant women who had history of blood transfusion (within the previous 2 weeks)
* Had any medical diseases
* Had risk pregnancy including bleeding disorders with multiple gestation Those who refused to consent

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 151 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
The degree of the adherence to the medication | at 28 and 36 weeks gestation
  Counting the total numbers of pills have been received (i.e. The numbers of dosage units (pills) that have been taken between two scheduled appointments were counted). Adherence to the supplementation regimen was calculated on the basis of the number of capsules remaining in the package at each return visit; adherence (%)=[30-number of pills left in the package/number of days between dispensing date and return date] ×100.

SECONDARY OUTCOMES:
Laboratory investigation for hemoglobin & ferrtin level | at 24 and 36 weeks gestation
  A sample of blood is tested in a lab. that helps to check the level of red blood cells (RBCs) and hemoglobin (Hb) concentration.
IRON Intake Calculation-Food Frequency Questionnaire (IRONIC-FFQ) | at 28 and 36 weeks gestation
  It was based on an iron food frequency assessment.All food products were categorized into twelve groups and thirty two related sub-groups characterized by a similar range of iron content. It consisted of open ended questions that specified the exact number of the individual consumption of iron food products during a typical week. To calculate the daily number of servings, the number of servings was divided by seven. The iron intake from the products was estimated by multiplying the daily number of servings by the typical iron content in one serving. A correlation coefficient was more than 0.85. Both in the assessment of validity and of reproducibility, a Bland-Altman index of 6.7% was recorded (93.3% of compared pairs of results were in the acceptable range, attributed to differences within ± 2 SD limit).
4) Dietary record diary (DRD). | at 28 and 36 weeks gestation
  It is self-record, an open-ended assessment method where the woman records all the foods and beverages consumed over a specific period of time thus minimizes reliance on memory

CONTACTS AND LOCATIONS:
Overall Officials: Rania Mahmoud A Ghani, PhD, Principal Investigator — Cairo University
Locations (1):
- Rania Mahmoud Abdel Ghani, Faisal, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rania MA. Effect of an Integrated Educational Session on Enhancing Compliance Behavior among Pregnant Women with Iron Deficiency Anemia. hptt//researchgate.com